CLINICAL TRIAL: NCT00236184
Title: E3810-A001-313: Efficacy and Safety of 10 mg Rabeprazole for Treating Heartburn in Frequent Sufferers
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Yufang Lu, Study Director, Eisai Medical Research Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E3810-A001-313
Record Dates: First submitted 2005-10-10; First posted 2005-10-12 (Estimated); Results first posted 2009-10-01 (Estimated); Last update posted 2010-04-06 (Estimated); Status verified 2010-03

CONDITIONS: Heartburn
MeSH Terms: conditions — Heartburn | interventions — Rabeprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Oral placebo tablet
  Interventions: Other: Placebo
- Rabeprazole sodium 10 mg (Experimental): oral rabeprazole 10 mg enteric-coated tablet
  Interventions: Drug: rabeprazole sodium

INTERVENTIONS:
Drug: rabeprazole sodium — Following a one week single-blind, placebo run-in phase, patients will receive rabeprazole 10 mg orally, once daily, for 14 days during the double-blind, randomized treatment phase. This will be followed by a one week single-blind placebo follow-up phase.
  Other Names: Aciphex
  Arms: Rabeprazole sodium 10 mg
Other: Placebo — Following a one week single-blind, placebo run-in phase, patients will receive placebo orally, once daily, for 14 days during the double-blind, randomized treatment phase. This will be followed by a one week single-blind placebo follow-up phase.
  Arms: Placebo

SUMMARY:
The purpose of this study is to investigate the safety and efficacy of rabeprazole sodium 10 mg in treating frequent heartburn.

DETAILED DESCRIPTION:
This is a multicenter, double-blind, randomized, placebo-controlled study to investigate the safety and efficacy of rabeprazole 10 mg in treating frequent heartburn. The study will last for up to five weeks and consists of the following three phases: a one to two week screening period that includes a one-week, single-blind, placebo run-in phase, a two week double-blind, randomized treatment phase, and a one week single-blind, placebo follow-up phase.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients > 18 years of age.
2. If female, not of childbearing potential by reason of surgery or menopause, or of childbearing potential, but using an approved method of contraception since the last menstrual period. Females of childbearing potential must have a negative serum pregnancy test before starting the study.
3. Patients must report a history of heartburn at least two days per week over the past month.

Exclusion Criteria:

1. History of erosive esophagitis verified by endoscopy.
2. History of gastroesophageal reflux disease (GERD) diagnosed by a physician.
3. Patients who have a history of Barrett's esophagus or esophageal stricture.
4. Evidence of any medical condition that may interfere with the conduct of the study, the interpretation of study results, or the health of the patient during the study.
5. Patients who require continuous use of proton pump inhibitors, histamine receptor (H2) blockers, or prokinetics. Prior intermittent use of these agents is permitted if they are discontinued at least three days prior to the run-in phase. The H2 blocker, cimetidine (Tagamet®), must be discontinued for at least seven days before the study drug is administered.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 629 (Actual)
Dates: Start 2005-10; Primary Completion 2006-03 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yufang Lu, MD, PhD, Study Director — Eisai Inc.
Locations (1):
- Jeffrey L. Newman, Vista, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was recruited at 39 centers in the US during the period of 10-Oct-2005 and 16-Mar-2006.
Pre-assignment Details: The screening phase (1 to 2 weeks) included a 1-week single-blind placebo run-in phase in order to determine baseline heartburn frequency and diary compliance. At the end of the run-in phase, subjects continued the study and entered the randomized treatment phase if they meet the study criteria.
Period: Overall Study
Arm/Group | Placebo | Rabeprazole 10 mg
Started | 310 | 319
Completed | 292 | 308
Not Completed | 18 | 11
Not completed — Adverse Event | 5 | 2
Not completed — Lack of Efficacy | 0 | 1
Not completed — Lost to Follow-up | 3 | 4
Not completed — Physician Decision | 1 | 1
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Protocol Violation | 3 | 0
Not completed — non-compliance with study drug | 2 | 1
Not completed — other | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Rabeprazole 10 mg: oral enteric-coated tablet
- Total: Total of all reporting groups
Arm/Group | Placebo | Rabeprazole 10 mg | Total
Number analyzed (Participants) | 310 | 319 | 629
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 285 | 298 | 583
  >=65 years | 25 | 21 | 46
Age Continuous [Mean (Standard Deviation); unit: years] | 45.4 (13.3) | 44.1 (14.4) | 44.7 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 198 | 186 | 384
  Male | 112 | 133 | 245
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 2 | 4
  Asian | 4 | 5 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 25 | 31 | 56
  White | 236 | 248 | 484
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 43 | 33 | 76
Region of Enrollment [Number; unit: participants]
  United States | 310 | 319 | 629

OUTCOME MEASURES:

1. Secondary Outcome: Summary of Percentage of Heartburn-free Daytimes, Intent-to-Treat (ITT) Population
Description: comparison between placebo and treatment will be analyzed using two-sample t-test.
Time Frame: 14-day treatment period.
Reporting Status: Not Posted
Measure: Mean (Standard Deviation); unit: Percentage of participants

2. Secondary Outcome: Summary of Percentage of Heartburn-Free Nighttimes,Intent-to-Treat (ITT) Population
Description: comparison between placebo and treatment will be analyzed using two-sample t-test.
Time Frame: 14-day treatment period.
Reporting Status: Not Posted
Measure: Mean (Standard Deviation); unit: Percentage of participants

3. Secondary Outcome: Change From Baseline in Average Regurgitation Severity Score Between Placebo and Rabeprazole.
Description: comparison between placebo and treatment will be analyzed using two-sample t-test.
Time Frame: 14-day treatment period.
Reporting Status: Not Posted
Measure: Mean (Standard Deviation)

4. Secondary Outcome: Change From Baseline in Average Belching Severity Score Between Placebo and Rabeprazole.
Description: comparison between placebo and treatment will be analyzed using two-sample t-test.
Time Frame: 14-day treatment period.
Reporting Status: Not Posted
Measure: Mean (Standard Deviation)

5. Primary Outcome: Complete Heartburn Relief During the First Full 24-Hour Period in the ITT Population.
Description: Subject was considered "complete relief" if he/she did not heartburn during the nighttime of the first dose date and no heartburn during the daytime of 1 day after the first dose date. The difference in complete relief within the first 24 hours between treatment groups was tested using a continuity corrected chi-square test without adjustment baseline heartburn severity.
Time Frame: first 24 hours
Population: The primary analysis will be on the intent-to-treat (ITT)population. ITT population includes all randomized subjects who received at least one dose of study drug and had at least one post-baseline assessment.
Measure: Number; unit: participants
Arm/Group | Placebo | Rabeprazole 10 mg
Number analyzed (Participants) | 306 | 318
participants | 114 | 163
Statistical Analysis 1: Comparison: Placebo vs Rabeprazole 10 mg; Test type: Superiority or Other; p < 0.001, Chi-squared, Corrected

ADVERSE EVENTS:
Arm/Group | Placebo | Rabeprazole 10 mg
Serious Adverse Events (participants affected / at risk) | 2/310 | 1/319
Other Adverse Events (participants affected / at risk) | 4/310 | 7/319
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=310) | Rabeprazole 10 mg (N=319)
Appendicitis perforated (Gastrointestinal disorders) | 1 (1) | 0 (0)
abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Chest pain (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=310) | Rabeprazole 10 mg (N=319)
Nasopharyngitis (Infections and infestations) | 4 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other